CLINICAL TRIAL: NCT06994819
Title: Double-blind Randomized Controlled Clinical Trial Under Dermatological Monitoring on Skin Tolerability and Efficacy of the Niostem Headset on Hair Growth, Hair Loss and Hair Quality After 3 and 6 Months of Daily Use
Brief Title: Evaluation of the Niostem Headset for Hair Growth and Hair Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mane Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ManeNio1.0
Record Dates: First submitted 2025-05-07; First posted 2025-05-29 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Androgenetic Alopecia; Pattern Baldness
Keywords: Hair loss; Alopecia; Androgenetic alopecia; Hair growth; Hair density; Hair quality; Niostem headset; Transcutaneous stimulation; Dermatology; Home-use device; Scalp stimulation; Non-invasive treatment; Clinical trial; Pattern baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: This was a parallel assignment study in which participants were randomly assigned to either the active niostem headset group or a placebo group. Both groups used their assigned device daily for 30 minutes over a period of 6 months. The study was conducted under double-blind conditions to evaluate skin tolerability and efficacy in reducing hair loss and promoting hair growth.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design: Participants, care providers, investigators, and outcome assessors were blinded to the assignment of active or placebo devices. The placebo devices visually resembled the active devices but did not deliver stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: niostem Headset (Experimental): Participants in this arm received the active niostem headset, a wearable electronic device designed to reduce hair loss and improve hair growth and quality. The device was applied once daily for 30 minutes over a 6-month period. Stimulation was administered through scalp-contact brush electrodes activated via a connected app.
  Interventions: Device: niostem headset (Active)
- Placebo Comparator: Sham Headset (Experimental): Participants in this arm received a placebo version of the niostem headset, which looked identical to the active device but did not deliver electrical stimulation. The sham device was worn once daily for 30 minutes over a 6-month period. This allowed the study to remain double-blind and helped assess the true efficacy of the active intervention.
  Interventions: Device: Sham niostem headset (Placebo)

INTERVENTIONS:
Device: niostem headset (Active) — The niostem headset is a non-invasive electronic stimulation device designed to reduce hair loss and improve hair growth. It delivers low-level electrical stimulation through brush electrodes that contact the scalp. Used once daily for 30 minutes for 6 months. Sessions are guided via a smartphone app.
  Arms: Active Comparator: niostem Headset
Device: Sham niostem headset (Placebo) — he sham niostem headset is visually identical to the active device but does not deliver electrical stimulation. Used once daily for 30 minutes for 6 months. Allows for blinding and placebo-controlled comparison.
  Arms: Placebo Comparator: Sham Headset

SUMMARY:
This double-blind, randomized, placebo-controlled clinical trial evaluates the Niostem headset, an electronic device designed to support hair growth, reduce hair loss, and improve hair quality. A total of 101 adult participants (20 female, 81 male) aged 18-55 were enrolled. Participants used the device daily for 30 minutes over a six-month period. The primary objective is to assess skin tolerability, and secondary objectives include evaluating usability and efficacy through validated questionnaires, TrichoScan hair analysis, and digital imaging under dermatological supervision.

DETAILED DESCRIPTION:
The study is conducted by Dermatest GmbH from October 2023 to September 2024 under dermatological supervision. The Niostem headset is a home-use electronic device applied daily for 30 minutes following standardized protocols. The primary endpoint is skin tolerability, with secondary endpoints assessing usability and potential effects on hair quality and growth.

Dermatological evaluations occur at baseline, 3 months, and 6 months. Quantitative assessments include TrichoScan imaging and digital macro photography, while subjective feedback is collected using validated self-report questionnaires. Participants are adults experiencing pattern hair loss-classified as Norwood stages 2-5 (men) and Ludwig stages I-II (women). Exclusion criteria include scalp conditions, pregnancy, ongoing medication use, and dermatological or psychiatric disorders. The study aims to assess the safety and user experience of a non-chemical, wearable neuromodulation device for cosmetic scalp and hair applications.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female volunteers between 18 and 55 years of age

Dermatologically confirmed pattern hair loss (Norwood stages 2-5 for men; Ludwig stages I-II for women)

Willingness to comply with daily use of the niostem headset for 6 months

No relevant scalp or dermatologic disease at baseline

Signed informed consent

Exclusion Criteria:

Scalp conditions (e.g., psoriasis, eczema, dermatitis)

Use of topical or systemic hair growth treatments within 3 months prior to study

Pregnancy or breastfeeding

Diagnosed psychiatric or neurologic disorders

Participation in another clinical study in the past 30 days

Known allergy to electrode gel or materials in the device

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Dermatological Adverse Reactions | Baseline, 3 months, and 6 months
  Assessment of skin tolerability via dermatological examination, identifying signs such as redness, irritation, pressure marks, or itching. Clinical assessments performed at each visit.

SECONDARY OUTCOMES:
Change in Hair Density (TrichoScan) | Baseline, 3 months, and 6 months
  Hair density measured in a defined scalp region using TrichoScan HD. Measurement area standardized per participant.
  Unit of Measure: Hairs per cm²
Change in Percentage of Anagen and Telogen Hairs | Baseline, 3 months, and 6 months
  Proportion of anagen-phase and telogen-phase hairs in the target area measured using TrichoScan HD.
  Unit of Measure: Percentage
Change in Percentage of Total, Terminal and Vellus Hairs | Baseline, 3 months, 6 months
  Total, Terminal and Vellus hair percentage evaluated in the defined target zone using TrichoScan HD.
  Unit of Measure: Percentage
Change in Global Scalp Hair Coverage (Photography) | Baseline, 3 months, and 6 months
  Standardized macro photographs taken at baseline and 24 weeks, evaluated for visual changes in overall hair coverage.
  Unit of Measure: Visual photographic comparison (qualitative assessment)
Participant-Reported Satisfaction with Hair Appearance, Comfort During Use and Perceived Efficacy | Baseline, 3 months, and 6 months
  Self-reported satisfaction scores, comfort levels and participants' perception of effectiveness in hair regrowth through standardized questionnaires.
  Unit of Measure: Score on a structured Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatest GmbH, Münster, NRW (Nordrhein-Westfalen), Germany

IPD SHARING:
Plan to Share IPD: No
The results of the clinical study will be published in a peer-reviewed journal. However, individual participant data (IPD) will not be shared due to privacy concerns and the proprietary nature of the device. Summary-level findings will be made publicly available through publication and clinical trial registry updates.

REFERENCES:
- [Background] Jellard S, Moore S, Chacon-Martinez CA. Novel Electrotrichogenic Device Promotes Hair Growth in Men With Androgenetic Alopecia: A Pilot Study. J Cosmet Dermatol. 2025 May;24(5):e70202. doi: 10.1111/jocd.70202. PMID 40296533